CLINICAL TRIAL: NCT05915663
Title: Impact of the Choice of Gastric Tube Placement Sites on the Incidence of Ventilator Associated Pneumonia and Other Complications in the Intensive Care Unit
Brief Title: Impact of the Choice of Gastric Tube Placement Sites on the Incidence of Ventilator Associated Pneumonia
Acronym: SONG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHM-2022/S03/05
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Intubated Patient Requiring a Gastric Tube
Keywords: orogastric tube; nasogastric tube; Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: Randomised cluster and cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasogastric (Experimental): nasogastric tube in period 1 and orogastric tube in period 2
  Interventions: Other: nasogastric tube and orogastric tube
- Orogastric (Experimental): orogastric tube in period 1 and nasogastric tube in period 2
  Interventions: Other: orogastric tube and nasogastric tube

INTERVENTIONS:
Other: nasogastric tube and orogastric tube — nasogastric tube in period 1 and orogastric tube in period 2
  Arms: Nasogastric
Other: orogastric tube and nasogastric tube — orogastric tube in period 1 and nasogastric tube in period 2
  Arms: Orogastric

SUMMARY:
In intensive care, many gastric tubes are inserted on a regular basis. There are different practices in terms of the location of the gastric tube. In some cases, the tube is inserted through the nose and in others, it is inserted through the mouth.

In the literature and in practice, these gastric tubes create discomfort and complications that have an impact not only on the patient, but also on the treatments and the length of the patient's stay in hospital.

Nosocomial Ventilator Associated Pneumonia is the most serious common complication for patients intubated with a gastric tube. It is possible that placement site may have an impact on the risk of developing Ventilator Associated Pneumonia, particularly by increasing the risk of bacterial pullulation opposite the sinuses when the tube is placed via the nasal route.

Investigator hypothesises that placing the gastric tube orally will reduce the rate of ventilator-associated pneumonia compared with the nasal route in mechanically ventilated intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* patient in intensive care, intubated, ventilated
* Adult
* Requiring a gastric tube
* With an expected duration of mechanical ventilation of more than 48 hours
* Affiliated to social security
* Patient or relative consent or, failing that, emergency inclusion of the patient

Exclusion Criteria:

* Pregnant, breast-feeding or parturient women
* Patients under legal protection: curatorship and guardianship
* Contraindication to placing a gastric tube through the nose or mouth
* Patients who already have a gastric tube when they enter the service
* Patient intubated for more than 24 hours
* Patient intubated via the nasotracheal route

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Compare impact of insertion site of gastric tube on the incidence of ventilator associated pneumoniae | Day 28
  The impact is measured by the number of ventilator associated peumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

REFERENCES:
- [Derived] Saletes J, Guitton C, Valleroy J, Guillarme S, Haubertin C, Paris G, Muller L, Rousseau C, Gamon P, L'Hotellier S, Forel JM, Roussel C, Garin A, Morand C, Maury E, Mangeard N, Menard L, Arnaud PY, Lejeune A, Rouanet E, Callahan JC. Effect of nasogastric versus orogastric tube placement on ventilator-associated pneumonia incidence in critically ill patients: a study protocol for a cluster randomised crossover trial in 16 intensive care units in France (SONG trial). BMJ Open. 2025 Sep 8;15(9):e099840. doi: 10.1136/bmjopen-2025-099840. PMID 40921641